CLINICAL TRIAL: NCT03306576
Title: Clinical Evaluation of Restorations Made of ELS Versus ELS Extra Resin Composite: A Prospective Randomized Controlled Clinical Trial up to 3 Years
Brief Title: Clinical Evaluation of ELS Versus ELS Extra Resin Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Saremco (Unknown)
Responsible Party: Principal Investigator, Funda Ozturk Bozkurt, DDS, PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.21426
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Caries, Dental
Keywords: composite restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Each participant will receive 2 matched restorations, one of each material.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ELS Extra composite (Experimental): Commercially available composite resin restorative that will be used for direct restoration as per manufacturer's instructions
  Interventions: Device: ELS Extra composite
- ELS composite (Active Comparator): Commercially available composite resin restorative that will be used for direct restoration as per manufacturer's instructions
  Interventions: Device: ELS composite

INTERVENTIONS:
Device: ELS Extra composite — One of the teeth will be restored using ELS composite. Procedures will be done under local anesthesia if necessary. The preparation and restoration of the tooth will be done according to to the guidelines for ordinary restorative techniques.
  Arms: ELS Extra composite
Device: ELS composite — the other teeth will be restored with a ELS resin composite with ordinary restorative techniques.
  Arms: ELS composite

SUMMARY:
Adhesive restorative materials are routinely used in operative dentistry to improve tooth tissues with minimal preparation, achieve more esthetic and long term restorations. Despite these efficacy to dentistry these materials still present some drawbacks like polymerization shrinkage. Postoperative sensitivity, marginal discoloration and possibly secondary caries are often associated with loss of marginal integrity in composite restorations occurred as a result of polymerization shrinkage. To achieve optimal long term performance, the requirements will be first to manage polymerization stress buildup following restoration.Low-shrinking composites with new formulas have been successful in brilliantly further developing the leader product els extra low shrinkage.

The objective of this controlled clinical trial is to evaluate the clinical performance of restorative material ELS versus ELS Extra resin composite for Class I and Class II cavities that needs to be restored in permanent teeth.

DETAILED DESCRIPTION:
The detrimental impact of resin composite polymerization shrinkage on restoration interface quality and stability has been recognized since the early use of this material is still one of the major drawbacks in adhesive dentistry, as it frequently leads to loss of marginal integrity or enamel fracture. According to clinical studies, drawbacks such as postoperative sensitivity, marginal discoloration and possibly secondary caries are often associated with loss of marginal integrity in composite restorations occurred as a result of polymerization shrinkage. Various technological solutions were investigated, including improved filler technology; improved, novel matrix structure with reduced shrinkage; use of stress-decreasing compounds within the resin matrix; changes in light-initiation technology to increase curing depth; and use of sonic vibrations and energy to favor flow and adaptation of highly filled resin composite. To achieve optimal long term performance, the requirements will be first to manage polymerization stress buildup following restoration. Low-shrinking composites should help to avoid clinical problems that are commonly associated with composite restorations, such as post-operative sensitivity, enamel cracks, rapid discoloration and deterioration of restoration margins, early development of caries recurrence, with a new formula and improved sculptability SAREMCO has been successful in brilliantly further developing the leader product els extra low shrinkage. When using new simplified restorative systems featuring distinctive physicochemical characteristics, the potential impact of different parameters such as fatigue behavior and/or elastic modulus on restoration quality and behavior is unknown and justifies additional investigations. Instead of in vitro evaluations, consideration of a rather well-established clinical trials suggesting medium to long term observation periods to discriminately appraise the clinical performance of various operative protocols.

The project includes 30 patients. Most of the patients have been recruited from the Istanbul Medipol University Dental Clinics in Istanbul. After giving their consent to take part in the study Class I & II restorations of both upper and lower molars and premolars are performed.The treatment procedure is: The patients are offered local anesthetic before treatment start. The cavity is excavated and filled according to the guidelines for composite restorations.

The control procedure is:

The restoration is evaluated according to marginal adaptation, cavo surface marginal discoloration, approximal contact, fractures, caries associated with restorations and postoperative hypersensitivity. The controls will take place after two weeks, one year, two years and three years.

ELIGIBILITY:
Inclusion Criteria:

* Primary caries removal
* Class I & II restoration replacement
* No obvious untreated caries, dental health problems (regularly checked by a dentist)
* Good or moderate oral hygiene (plaque score of less than 30% in anterior region be-fore treatment)
* No untreated periodontal disease (only DPSI 1, 2)
* Subjects had to present no active carious lesions
* Subjects had to be over the age of 18, be classified according to the American Society of Anesthesiologists (ASA) as ASA I or ASA II, present with good oral hygiene, and be free of periodontal disease (probing depth and attachment levels within normal limits, no furcation involvement, and no mobility)
* Subjects had to agree to keep the scheduled recall appointments for data collection and maintenance and plan to stay in the area for at least 3 years.

Exclusion Criteria:

* Caries extends cemento-enamel junction in Class II.
* Considerable horizontal and/or vertical mobility of teeth: tooth mobility index score 2 or 3
* Considerable periodontal disease without treatment (DPSI 3-, 3+ and 4)
* Endodontic treatment with extensive loss of tooth tissue
* Patients who still want to bleach their teeth or bleached teeth less than 3 weeks ago
* Excluding the teeth, with opposing natural dentition (either intact or restored with intracoronal or extracoronal fixed restorations), and with a minimum of 20 teeth
* Subjects who presented with severe wear facets and/or reported parafunctional activities such as clenching or nocturnal bruxism
* Subjects who were restored with a removable partial dental prosthesis (RPDP), unless the RPDP replaced the tooth that was planned to be restored in the study
* Subjects who were pregnant pregnant during the duration of the study
* Subjects who are known to be allergic to the ingredients of resin materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Modified FDI criteria | 3 years
  Restoration failure is based on clinical performance criteria according to the modified FDI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Mutlu Ozcan, Prof Dr,PhD, Principal Investigator — University of Zurich, Center for Dental Materials Unit, Center for Fixed and Removable Prosthodontics and Dental Materials Science
Locations (1):
- Istanbul Medipol University, Dental School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No